CLINICAL TRIAL: NCT06267547
Title: Healthy Activities Improve Lives Randomized Control Trial
Brief Title: Healthy Activities Improve Lives (HAIL)
Acronym: HAIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Associate Director and Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P003522
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIL Online Platform + Fit and Strong! Program (Experimental): Participants (N=60) will be recruited from two racially diverse churches or senior centers (30 participants per church/center) to examine the efficacy of the HAIL Online platform + F&S! program for older adults in black communities. Participants will complete the 8-week F&S! exercise program (with access to the adjunct HAIL online platform), which will be delivered in-person as well as remote, and then continue to use the HAIL online platform during the 3-mo follow-up.
  Interventions: Other: HAIL Online Platform; Behavioral: Fit and Strong! Program
- Fit and Strong! Program (Active Comparator): Participants (N=60) will be recruited from two racially diverse churches or senior centers (30 participants per church/center) to examine the feasibility and acceptability of the HAIL Online platform. Participants will complete the 8-week F&S! exercise program (without access to the adjunct HAIL online platform), which will be delivered in-person as well as remote, and then complete the 3-mo follow-up.
  Interventions: Behavioral: Fit and Strong! Program

INTERVENTIONS:
Other: HAIL Online Platform — The HAIL online platform was developed based on feedback from our focus groups with older adults affiliated with BMA churches (conducted per IRB Protocol 2020P003100). Specifically, the HAIL online platform has a landing page where participants can access the links to the F&S! exercise sessions, complete the exercise log, obtain tips from an exercise instructor, as well as view study announcements. The landing page has a navigation bar on the left to access 1) the study assessments; 2) the F&S! exercise program participant manual; and 3) information on how to contact study staff. The goal of this adjunctive HAIL online platform is to support the continuation of exercise in the follow-up period once the 8-week F&S! exercise program is over. We conducted an open trial (per IRB protocol 2022P001782) to assess the feasibility and acceptability of the HAIL online platform adjunct to the F&S! program, which yielded positive results.
  Arms: HAIL Online Platform + Fit and Strong! Program
Behavioral: Fit and Strong! Program — The Fit and Strong! Program (F&S!) is an exercise program for older adults developed by a study consultant, Dr. Susan Hughes, with funding from the National Institute of Aging. It is tailored for the unique needs of older, underserved adults and targets modifiable factors depicted by the socioecological model is necessary. The F&S! exercise program assists older adults to improve strength and functioning.

SUMMARY:
The investigators have developed an online platform to support the 8-week, F&S! exercise program called the Healthy Activity Improves Lives (HAIL) online platform. The aim of this study is to perform a cluster randomization of four racially diverse churches or senior centers to either the standard F&S! program, or the combined HAIL Online Platform + F&S! program to examine the efficacy of the HAIL online platform + F&S! program for older adults in black communities.

DETAILED DESCRIPTION:
This is randomized clinical trial of cluster randomization evaluating the efficacy and feasibility of the HAIL online platform + F&S! program. We will enroll four cohorts (i.e., at two racially diverse churches or senior centers) for a total number of 120 participants. We will use a phone screen to assess participants' eligibility and explain the study procedures. Eligible individuals will then be given a link to complete an e-Consent in REDCap. Those randomized into the intervention group will also receive instructions on how to access the HAIL online platform to complete assessments as part of the baseline visit. Participants in both the intervention and comparison groups will complete the 8-week F&S! exercise program which will be delivered in-person as well as remote. Participants in the intervention group will have access to the adjunct HAIL online platform during the F&S! program, and then continue to use the HAIL online platform during the 3-mo follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 55 years
* Participants are able to travel to one of the churches for the in-person F&S! exercise sessions
* Participants cannot be currently participating in a regular PA program (i.e., at least 100 min per week of moderate to vigorous physical activities)

Exclusion Criteria:

* Participants do not understand study procedures or are unable to participate in the verbal consent process
* Participants must have a physician responsible for their medical care
* Participants endorse an item on the Revised Physical Activity Readiness Questionnaire (rPAR-Q) as confirmed by their treating physician
* Participants who report any contraindication to exercising (e.g., recent ECG changes or myocardial infarction, unstable angina, uncontrolled arrhythmias, third degree heart block, congestive heart failure)
* Participants who receive a score of 28 or higher on the Telephone Interview for Cognitive Status (TICS) during pre-screening

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Retention | Week 20
  Retention will be assessed by how many individuals completed the 3-month post-intervention follow-up
Acceptability | Week 8
  Acceptability will be assessed by the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 assesses acceptability and feasibility of the HAIL online platform and has demonstrated good reliability and validity. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Acceptability (Feedback Form) | Week 20
  Acceptability will be assessed by the HAIL online Feedback form. We will develop a form to ask for tailored feedback on the F&S! program and the HAIL online platform to better understand participants' satisfaction with specific aspects of this online program.
Acceptability (Exit Interviews) | Week 20
  Acceptability will finally be assessed with focus group exit interviews, which will be qualitatively coded.

SECONDARY OUTCOMES:
Changes in Physical Activity (Steps) | Weeks 0, 8, 20
  Changes in physical activity will be measured by Participants' daily step counts. This outcome will be measured via the GT3X ActiGraph accelerometer.
Changes in Physical Activity (MVPA) | Weeks 0, 8, 20
  Changes in physical activity will be measured by participants' daily number of minutes of moderate to vigorous physical activity (MVPA). This outcome will be measured via the GT3X ActiGraph accelerometer.
Changes in Aerobic Capacity | Weeks 0, 8, 20
  This outcome will be measured via the 6 minute Walk Test.
Changes in Physical Strength | Weeks 0, 8, 20
  This outcome will be measured via the Timed-Stands Test.
Motivation to Change | Week 0
  Motivation to change outcome will be measured via the Readiness for Change Form. This is used to measure participants' motivation to participate in exercising. A high score indicates the respondent is more interested in participating in exercise activities. A low score indicates the respondent is less interested in participating in exercise activities.
Utilization of Healthcare Resources | Week 0
  Utilization of healthcare resources outcome will be assessed via the Healthcare Utilization Form. This a descriptive measure used to assess utilization of healthcare resources in the past 6 months, and to better characterize the sample based on the number of comorbid conditions present. There is no scoring or total score.
Fall History | Week 0
  Fall history outcome will be measured via the Fall History Form. This form is used to assess the history of falling within the past two years in participants.
Chronic Conditions | Week 0
  Chronic conditions outcome will be measured via the Geri-AIMS. This is a19-item self-administered questionnaire adapted from the Arthritis Impact Measurement Scales (AIMS) for use with frail elderly respondents. The questionnaire assesses the presence of existing chronic medical conditions.
Changes in Overall Wellbeing | Weeks 0, 8, 20
  Wellbeing will be measured via the WHO(Five) Well-Being Index (WHO-5). This is a reliable psychometric measure that predicts depression. The questionnaire consists of five items that assess predictors of depressive symptoms: positive mood, energy and interest. The raw score is calculated by totaling the figures of the five answers. The raw score ranges from 0 to 25, 0 representing worst possible and 25 representing best possible quality of life.
Changes in Depression | Weeks 0, 8, 20
  Depression outcome will be measured via the Patient Health Questionnaire (PHQ-9). This is a 9-item, standardized and validated questionnaire that assesses the prevalence and severity of depression based on the DSM-5 criteria. The raw score ranges from 0 to 27, 1 representing minimal depression and 27 representing severe depression.
Changes in Anxiety | Weeks 0, 8, 20
  Anxiety outcome will be measured via the Generalized Anxiety Disorder 7-item (GAD-7) scale. This is a 7-item anxiety scale with good reliability, as well as criterion, construct, factorial, and procedural validity. The raw score ranges from 0 to 21. Increasing scores are associated with multiple domains of functional impairment. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Changes in Physical Functioning | Weeks 0, 8, 20
  Physical function outcome will be measured via the Patient-Reported Outcomes Measurement Information-Physical Functiong. This is an 8-item scale assessing coordination, functional mobility, strength and upper extremity function. The raw score ranges from 0 to 40. Increasing scores are associated with higher physical functioning.
Changes in Social Isolation | Weeks 0, 8, 20
  Social isolation outcome will be measured via the Patient-Reported Outcomes Measurement Information Short Form- Social Isolation 4. This is a 4-item scale used to capture participants' perception of being left out and disconnected from others. The raw score ranges from 0 to 20. Increasing scores are associated with higher feelings of social isolation.
Changes in Confidence in Exercises | Weeks 0, 8, 20
  Exercise confidence outcome will be measured via the Exercise Confidence Form. This is a 4-item questionnaire used to assess confidence in doing certain physical activities. The raw score ranges from 0 to 40. Increasing scores are associated with higher confidence in exercise.

OTHER OUTCOMES:
Satisfaction with program | Week 8
  This outcome will be measured via the Client Satisfaction Questionnaire (CSQ-8). Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Satisfaction with program | Week 20
  This outcome will be measured via the Client Satisfaction Questionnaire (CSQ-8). Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Use of online program | Week 8
  This outcome will be assessed via the F&S! Program feedback from. This form consists of 8 questions and a semistructured exit interview of 4 questions. There is no scoring or total score.
Use of online program | Week 20
  This outcome will be assessed via the F&S! Program feedback from. This form consists of 8 questions and a semistructured exit interview of 4 questions. There is no scoring or total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Roslindale Baptist Church, Boston, Massachusetts, United States